CLINICAL TRIAL: NCT02532465
Title: Glottic View Using Supraglottic Devices in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Senthil G. Krishna (Other)
Responsible Party: Sponsor-Investigator, Senthil G. Krishna, Assistant Clinical Professor, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB15-00486
Record Dates: First submitted 2015-08-21; First posted 2015-08-25 (Estimated); Results first posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-07

CONDITIONS: Operative Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Air-Q (Active Comparator): The Air-Q is composed of an airway tube that connects to an elliptical mask with a cuff which is inserted through the patient's mouth, down the windpipe, and once deployed forms an airtight seal on top the glottis (unlike tracheal tubes which pass through the glottis) allowing a secure airway to be managed by a health care provider.
  Interventions: Device: Air-Q
- i-gel (Experimental): The i-gel is designed to create a non-inflatable anatomical seal of the pharyngeal, laryngeal and perilaryngeal structures whilst avoiding the compression trauma that can occur with inflatable supraglottic airway devices.
  Interventions: Device: i-gel

INTERVENTIONS:
Device: Air-Q
  Arms: Air-Q
Device: i-gel
  Arms: i-gel

SUMMARY:
Endotracheal intubation is the gold standard for securing the airway. However, while managing patients with difficult airways, various supraglottic devices have been used as rescue airway devices. The aim of this study is to compare the fiberoptic view through the internal aspect of the i-gel versus the Air-Q LMA in pediatric patients. By examining the fiberoptic view through these two devices, the investigators will determine which device provides a clearer passage to the glottic opening and is therefore the preferred conduit to aid endotracheal intubation in difficult airways.

ELIGIBILITY:
Inclusion Criteria:

* Patients less than 18 years of age who will be receiving an LMA as part of standard of care for their procedure.

Exclusion Criteria:

* None

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2015-08; Primary Completion 2018-07-26 (Actual); Study Completion 2018-09-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Air-Q: The Air-Q is composed of an airway tube that connects to an elliptical mask with a cuff which is inserted through the patient's mouth, down the windpipe, and once deployed forms an airtight seal on top the glottis (unlike tracheal tubes which pass through the glottis) allowing a secure airway to be managed by a health care provider.
  Air-Q
- I-gel: The i-gel is designed to create a non-inflatable anatomical seal of the pharyngeal, laryngeal and perilaryngeal structures whilst avoiding the compression trauma that can occur with inflatable supraglottic airway devices.
  i-gel
Period: Overall Study
Arm/Group | Air-Q | I-gel
Started | 25 | 25
Completed | 24 | 24
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Air-Q | I-gel | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 14 [6 to 16] | 12 [7 to 16] | 13 [7 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 12 | 10 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
Weight [Median (Inter-Quartile Range); unit: kilograms] | 50 [22 to 70] | 49 [26 to 69] | 49 [25 to 70]

OUTCOME MEASURES:

1. Primary Outcome: Acceptable View of the Glottic Aperature (Grade I-II)
Description: Grade I view - Glottic aperture seen completely without any obstruction, Grade II view - Glottic aperture seen only partially but visual obstruction is less than 50%.
Time Frame: 15 seconds after insertion of Air-Q or i-gel
Measure: Number; unit: participants
Arm/Group | Air-Q | I-gel
Number analyzed (Participants) | 24 | 24
participants | 20 | 21

2. Secondary Outcome: Airway Insertion Time
Description: Amount of time it takes to insert airway.
Time Frame: Immediately after anesthesia induction
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Air-Q | I-gel
Number analyzed (Participants) | 24 | 24
seconds | 19 [16 to 20] | 21 [16 to 29]

3. Secondary Outcome: Time to Achieve Best Fiberoptic View
Description: After confirmation of adequate placement and ventilation, a flexible fiberoptic bronchoscope was inserted through the stem of the supraglottic device to visualize the glottic aperture. The time taken for bronchoscopy, defined as time from disconnection of the anesthetic circuit from the SGA to first visualization of the glottic aperture, was recorded.
Time Frame: 15 seconds after insertion of Air-Q or i-gel
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Air-Q | I-gel
Number analyzed (Participants) | 24 | 24
seconds | 25 [20 to 30] | 21 [17 to 40]

ADVERSE EVENTS:
Time Frame: Day of surgery
Arm/Group | Air-Q | I-gel
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-07): https://cdn.clinicaltrials.gov/large-docs/65/NCT02532465/Prot_SAP_000.pdf